CLINICAL TRIAL: NCT03749720
Title: Can Digital Droplet PCR (ddPCR) on Blood Samples From Patients With HPV Related Cancers Become a Reality in Cancer Treatment and Monitoring?
Brief Title: HPV in Blood Samples From Cervical Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U416
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2021-09

CONDITIONS: HPV-Related Carcinoma; HPV-Related Malignancy
Keywords: Cervical Cancer; HPV; Pathology; ddPCR
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Case-control study with 141 case patients newly diagnosed cervical cancer and a control group of 10 healthy women with no prior cervical dysplasia and 25 women with cervical dysplasia (CIN3), respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical cancer patients (Other): Baseline- and follow-up blood samples are collected from the cervical cancer patients at time of diagnosis and during treatment and clinical follow-up. HPV DNA is measured in these samples.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample taken from cervical cancer patients at time of diagnosis (baseline) and follow-up visits.

SUMMARY:
By means of digital droplet PCR (ddPCR) anf targeted Next Generation Sequencing (NGS), this study examines blood samples from patients newly diagnosed with cervical cancer to investigate whether it is possible to measure the presence and amount of HPV DNA in these blood samples. The first blood sample is taken at time of diagnosis, and follow-up blood samples are collected during treatment- and follow-up visits. We expect to find a correlation between the disease stage and the viral load and also a decline in viral load after treatment. Furthermore, we hope that this method may serve as a way of detecting disease recurrence earlier than what is possible today.

DETAILED DESCRIPTION:
This study hypothesises that in patients with HPV-related cervical cancer, HPV DNA may be released into the bloodstream from tumor cells. These fragments of HPV DNA shed by tumor may therefore be measured in blood samples from the patients. By using the same setting as for real-time PCR with PCR primers and probes for fluorescence detection, the study uses digital droplet PCR (ddPCR), a method based on dilution and partitioning of the blood sample in many reaction chambers or droplets, to measure absolute quantities of HPV DNA fragments in blood samples from women with different stages of cervical cancer. Furthermore, our research group has developed in-house amplicon-based Next Generation Sequencing (NGS) assays for HPV detection and genotyping (the NGS HPV genotyping panel) and HPV integration status and variants (the HPV16 panel), and blood samples are also analysed with the NGS HPV genotyping panel. Cervical tissue samples from primary tumor are collected and analysed with the NGS HPV genotyping panel, and HPV16 positives are further analysed with the NGS HPV16 panel. Patients are recruited at the time of diagnosis, where a baseline blood sample is collected. Follow-up blood samples are collected during treatment and at follow-up visits up to two years after the diagnosis. We expect the HPV DNA load to decrease after treatment, and if an increase in viral load is detected during follow-up, we expect this to be an early sign of a disease recurrence. The method may therefore become an effective monitoring tool in these patients in terms of detecting a ongoing disease recurrence, which gives us the chance to intervene and treat these patients before the disease becomes too disseminated.

For included patients experiencing af recurrence of their disease, tissue samples from recurrent disease are collected and analysed with both the NGS HPV genotyping panel, the NGS HPV16 panel (for HPV16 positives), p16 staining, and a panel detecting relevant somatic mutations in the TP53 and RB1 tumor suppressor proteins.

ELIGIBILITY:
Inclusion Criteria cases:

* Diagnosed with cervical cancer ≥ stage 1B between june 2018 and june 2020
* > 18 years of age at the time of diagnosis
* There must be available cervical tissue material from the patient to analyse for HPV

Inclusion Criteria healthy controls

* Women > 18 years with no prior history of any cervical dysplasia

Inclusion Criteria CIN3 controls

* Women > 18 years
* Must have a histologically verified severe cervical dysplasia (CIN3)
* Is admitted for cervical conisation

Exclusion Criteria cases:

* < 18 years of age at time of cervical cancer diagnosis
* Cervical cancer < stage 1B

Exclusion Criteria healthy controls:

* < 18 years of age
* Prior cervical dysplasia

Exclusion Criteria CIN3 controls:

* < 18 years of age
* Women with only low grades of cervical dysplasia (CIN1 or CIN2)
* Women with HPV-negative cervical biopsies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
HPV DNA | Two years
  A qualitative and quantitative measure of HPV DNA in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bønløkke, MD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Obstetrics and Gynecology, Aarhus
  - Department of Obstetrics and Gynecolgy, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonlokke S, Stougaard M, Sorensen BS, Parner E, Nyvang GB, Lindegaard JC, Blaakaer J, Bertelsen J, Fuglsang K, Steiniche T. Ultrasensitive next-generation sequencing-based detection of circulating human papillomavirus DNA for cervical cancer recurrence monitoring. Cancer. 2026 Feb 15;132(4):e70282. doi: 10.1002/cncr.70282. PMID 41653072